CLINICAL TRIAL: NCT05475990
Title: Comparison of 6% Hydroxyethyl Starch (130/0.4) and Crystalloid Coload Combined With Prophylactic Norepinephrine Infusion for Postspinal Anesthesia Hypotension in Patients Undergoing Caesarean Section
Brief Title: Comparison of Hydroxyethyl Starch and Crystalloid Coload Combined With Norepinephrine Infusion for Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2022-3
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-07

CONDITIONS: Adverse Effect
Keywords: Crystalloid; Hydroxyethyl starch 130/0.4; Postspinal anesthesia hypotension; Cesarean section; Norepinephrine; Coload
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Colloids; Crystalloid Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxyethyl starch coload group (Experimental): 10 ml/kg 6% Hydroxyethyl starch (130/0.4) coload combined with an initial infusion dose of prophylactic norepinephrine simultaneous with spinal anesthesia
  Interventions: Drug: Hydroxyethyl starch
- Crystalloid coload group (Experimental): 10 ml/kg crystalloid coload combined with an initial infusion dose of prophylactic norepinephrine simultaneous with spinal anesthesia.
  Interventions: Drug: Crystalloid

INTERVENTIONS:
Drug: Hydroxyethyl starch — 10 ml/kg 6% Hydroxyethyl starch (130/0.4) coload combined with an initial infusion dose of prophylactic norepinephrine (0.025 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.005 ug/kg/min of prophylactic norepinephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Colloid
  Arms: Hydroxyethyl starch coload group
Drug: Crystalloid — 10 ml/kg crystalloid coload combined with an initial infusion dose of prophylactic norepinephrine (0.025 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.005 ug/kg/min of prophylactic norepinephrine according to the responses of previous patients according to the up-down sequential allocation.
  Arms: Crystalloid coload group

SUMMARY:
The purpose of this study is to investigate the ED50 and ED90 for an effective 6% Hydroxyethyl starch (130/0.4) or crystalloid coload combined with prophylactic norepinephrine infusion dose for postspinal anesthesia hypotension in patients undergoing cesarean section.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. Colloid fluid coload has been highly demonstrated for prevention and/or treatment of post-spinal anesthesia hypotension. In addition, there's some evidence that prophylactic infusion of norepinephrine could effectively reduce the incidence of post-spinal anesthesia hypotension in parturients undergoing cesarean section. However, the ED50 and ED90 for an effective 6% Hydroxyethyl starch (130/0.4) or crystalloid coload combined with prophylactic norepinephrine infusion dose for postspinal anesthesia hypotension is still unknown. The purpose of this study is to investigate the ED50 and ED90 for an effective 6% Hydroxyethyl starch (130/0.4) or crystalloid coload combined with prophylactic norepinephrine infusion dose for postspinal anesthesia hypotension in patients undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Primipara or multipara
* Singleton pregnancy ≥ 37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥ 160mmHg
* Hemoglobin < 7g/dl
* Coagulation or renal function disorders
* Known allergy to hydroxyethyl starch
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
ED 50 and ED 90 | 1-15 minutes after spinal anesthesia
  The dose of prophylactic norepinephrine combined with 10 ml/kg 6% Hydroxyethyl starch (130/0.4) or 10 ml/kg crystalloid coload that would be effective in preventing postspinal anesthesia hypotension in 50% (effective dose, ED 50) and 90% (ED90) of patients

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline.
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia
  Heart rate < 60 beats/min.
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery
  From umbilical arterial blood gases.
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases.
Base excess (BE) | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University; Xiangzhao Xu, M.D.; Ph. D, Study Chair — The People's Hospital of Nanchuan
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China